CLINICAL TRIAL: NCT03433625
Title: Behavioural Experiments for Intolerance of Uncertainty: A 6-session Treatment for Generalized Anxiety Disorder
Brief Title: 6-Session Treatment for Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Quebec en Outaouais (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Concordia University, Montreal (Other); University College, London (Other)
Responsible Party: Principal Investigator, Michel Dugas, Ph.D., Professor of Psychology, Universite du Quebec en Outaouais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2252
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: Cognitive-behavioural therapy
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioural experiments (CBT) (Experimental): Behavioural experiments involve selecting a specific thought to be tested (e.g., "uncertainty makes me unable to act") and designing a detailed experiment to test out the thought.
  Interventions: Behavioral: Behavioural experiments for intolerance of uncertainty (BE-IU)
- Waiting list (No Intervention): 6 week wait (with assessments) before being transferred to the experimental condition.

INTERVENTIONS:
Behavioral: Behavioural experiments for intolerance of uncertainty (BE-IU) — CBT
  Arms: Behavioural experiments (CBT)

SUMMARY:
Generalized Anxiety Disorder (GAD) is a chronic condition that is characterized by excessive and uncontrollable worry and anxiety. In Canada, 3 to 4% of the population suffer from GAD at any point in time. These individuals have a lowered quality of life and are at risk for many medical conditions such as coronary heart disease and cancer. Research suggests that both pharmacological and psychological approaches are effective for treating GAD in the short-term; however, psychological treatments appear to offer the greatest long-term benefits. There exist a number of effective psychological treatments for GAD, most of which fall into the category of cognitive-behavioural therapy or CBT. In the 1990s, a group of Canadian investigators developed a CBT protocol for GAD that included four components. Data from five clinical trials suggest that one of the four components is particularly important for treatment success: experiencing uncertainty rather than avoiding it in everyday life. Stated differently, learning to tolerate and deal with uncertainty appears to be the key to decreasing worry and anxiety. Given this finding, the investigators have developed a new treatment that exclusively targets intolerance of uncertainty: Behavioural Experiments for Intolerance of Uncertainty or BE-IU. The goal of the current proposal is to test the efficacy of BE-IU (6 weekly treatment sessions) by comparing it to a Waiting List (WL) control condition (6 weeks). A total of 50 participants with a primary diagnosis of GAD will be randomly assigned to either BE-IU or WL and will be assessed at 4 time points ranging from pre-treatment to 12-month follow-up. The conditions will be compared in terms of treatment efficacy and mechanisms. The investigators will also examine the predictors of change during the 12-months following treatment. The proposed study will produce data on the efficacy and mechanisms of a treatment for GAD that is less costly, less complex and easier to disseminate than treatments that are currently available.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age;
2. principal diagnosis of GAD;
3. no change in medication type or dose in 4 to 12 weeks before study entry (4 weeks for benzodiazepines, 12 weeks for antidepressants and hypnotics);
4. willingness to keep medication status stable while participating in the study;
5. no use of herbal products known to have CNS effects in the 2 weeks before study entry;
6. no evidence of suicidal intent (based on clinical judgement);
7. no evidence of current substance abuse, current or past schizophrenia, bipolar disorder or organic mental disorder;
8. no current participation in other trials;
9. no concurrent psychotherapy during treatment phase of trial;
10. no evidence of anxiety symptoms due to a general medical condition based on clinical judgement (e.g., clinical hyperthyroidism, hypoglycaemia, anaemia).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Clinician's Severity Rating (CSR) of Anxiety Disorders Interview Schedule (ADIS) | 8 weeks
  Structured diagnostic interview

SECONDARY OUTCOMES:
Penn State Worry Questionnaire | 8 weeks
  16-item self-report questionnaire measuring trait worry. Only the total score is reported (range: 16 to 80). Higher values represent a worse outcome.
Worry and Anxiety Questionnaire | 8 weeks
  11-item self-report questionnaire measuring diagnostic criteria for generalized anxiety disorder. Only the total score is reported (range: 7 to 35). Higher values represent a worse outcome.
Beck Anxiety Inventory | 8 weeks
  21-item self-report questionnaire measuring anxiety over the past week. Only the total score is reported (range: 0 to 63). Higher values represent a worse outcome.
Beck Depression Inventory-II | 8 weeks
  21-item self-report questionnaire measuring depressive symptoms over the past 2 weeks. Only the total score is reported (range: 0 to 63). Higher values represent a worse outcome.

OTHER OUTCOMES:
Intolerance of Uncertainty Scale | 8 weeks
  27-item self-report questionnaire measuring negative beliefs about uncertainty. Only the total score is reported (range: 27 to 135). Higher values represent a worse outcome.
Safety Behaviours Questionnaire | 8 weeks
  18-item self-report questionnaire measuring the use of avoidance and safety behaviors. Only the total score is reported (range: 18 to 90). Higher values represent a worse outcome.
Heart rate variability | 8 weeks
  Heart rate monitoring with chest strap and Polar watch
Acceptance and Action Questionnaire, second edition | 8 weeks
  10-item self-report questionnaire measuring acceptance of internal experiences and commitment to valued action. Only the total score is reported (range 10 to 70). Higher values represent a better outcome.
Pain Catastrophizing Scale | 8 weeks
  13-item self-report questionnaire measuring negative beliefs about pain. Only the total score is reported (range: 0 to 52). Higher values represent a worse outcome.
Agression Questionnaire | 8 weeks
  12-item self-report questionnaire measuring the tendency to become angry. Only the total score is reported (range: 12 to 60). Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michel J Dugas, Ph.D., Principal Investigator — Université du Québec en Outaouais
Locations (1):
- Universite du Quebec en Outaouais, Gatineau, Quebec, Canada